CLINICAL TRIAL: NCT03414294
Title: A Phase I Single-Center, Randomized, Double-Blind, Placebo-Controlled, Combined Single Ascending Dose, Multiple Ascending Dose, and Food Effect Study to Investigate the Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of K-755 in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Safety of K-755 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Company, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: K-755-1.01AU
Record Dates: First submitted 2018-01-09; First posted 2018-01-29 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Intervention Model Description: Sequential Assignment/Crossover (for food effect)
Who Masked: Participant, Investigator
Masking Description: Masking for Part A (SAD) , Part B (MAD), Part E (MAD) open for Part C (FE) and Part D (FE)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- K-755 Part A (SAD) (Experimental)
  Interventions: Drug: K-755 Part A (SAD)
- Placebo Part A (SAD) (Placebo Comparator)
  Interventions: Drug: Placebo Part A (SAD)
- K-755 Part B (MAD) (Experimental)
  Interventions: Drug: K-755 Part B (MAD)
- Placebo Part B (MAD) (Placebo Comparator)
  Interventions: Drug: Placebo Part B (MAD)
- K-755 Part C (FE) (Experimental)
  Interventions: Drug: K-755 Part C (FE)
- K-755 Part D (FE) (Experimental)
  Interventions: Drug: K-755 Part D (FE)
- K-755 Part E (MAD) (Experimental)
  Interventions: Drug: K-755 Part E (MAD)
- Placebo Part E (MAD) (Placebo Comparator)
  Interventions: Drug: Placebo Part E (MAD)

INTERVENTIONS:
Drug: K-755 Part A (SAD) — Single ascending dose (SAD). There will be 7 cohorts in the Part A. Three quarters of subjects will receive K-755 tablet orally in a double-blind fashion.
  Arms: K-755 Part A (SAD)
Drug: Placebo Part A (SAD) — Single ascending dose (SAD). In Part A, one quarter of subjects will receive placebo tablet orally in a double-blind fashion.
  Arms: Placebo Part A (SAD)
Drug: K-755 Part B (MAD) — Multiple ascending dose (MAD). There will be 4 cohorts in the Part B. Three quarters of subjects will receive K-755 oral tablet in a double-blind fashion.
  Arms: K-755 Part B (MAD)
Drug: Placebo Part B (MAD) — Multiple ascending dose (MAD). In Part B, one quarter of subjects will receive placebo tablet orally in a double-blind fashion.
  Arms: Placebo Part B (MAD)
Drug: K-755 Part C (FE) — Food effect (FE). All subjects in Part C will receive K-755 oral tablet both under fed and fasted condition in a open-label, crossover fashion.
  Arms: K-755 Part C (FE)
Drug: K-755 Part D (FE) — Food effect (FE). All subjects in Part D will receive K-755 oral tablet both under fed and fasted condition in a open-label, crossover fashion.
  Arms: K-755 Part D (FE)
Drug: K-755 Part E (MAD) — Multiple ascending dose (MAD). There will be 2 cohorts in the Part E. Three quarters of subjects will receive K-755 oral tablet in a double-blind fashion.
  Arms: K-755 Part E (MAD)
Drug: Placebo Part E (MAD) — Multiple ascending dose (MAD). In the Part E. One quarter of subjects will receive placebo tablet orally in a double-blind fashion.
  Arms: Placebo Part E (MAD)

SUMMARY:
This is a Phase 1 study designed to explore the safety, tolerability and pharmacokinetics of K-755 following oral administration to healthy male and female volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
2. Males or females, of any race, between 18 and 45 years of age.
3. Body mass index (BMI) between 18.0 and 28.0 kg/m2.
4. Hematology, clinical chemistry, and urinalysis test results within the reference ranges or showing no clinically relevant deviations, as judged by the Investigator.
5. No clinically significant abnormalities on the basis of medical history, physical examination findings, and vital signs.
6. All females must have a negative serum pregnancy test.
7. Able and willing to comply with the protocol and study procedures.

Exclusion Criteria:

1. Female subject who are pregnant or breastfeeding.
2. Subject with presence of active or recurring clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal, or metabolic disease requiring medical treatment.
3. Subject with any surgical or medical condition that might significantly alter the absorption, distribution, metabolism, or excretion of K-755.
4. Subject with presence of an active malignancy or within the past 5 years a malignancy of any type, other than basal cell carcinoma of the skin.
5. Subject has a history of type 1 hypersensitivity to any medication and/or clinically relevant food allergies.
6. Subject has a history of drug addiction.
7. Subject has a positive screen for drugs of abuse, cotinine or alcohol.
8. Subject has a history of regular alcohol consumption within 6 months of the study.
9. Subject has smoked tobacco within 6 months prior to Check-in, or has used non-inhaled tobacco- or nicotine-containing products within 3 months prior to Check-in.
10. Subject has used prescription or over-the-counter medications, dietary/nutritional supplements (except paracetamol or vitamin supplements)
11. Subject has used steroid medications (oral, inhaled, parenteral, or topical) within 30 days or 5 half-lives (whichever is longer) before study drug administration.
12. Subject has participated in an investigational drug study within 30 days or 5 half-lives (whichever is longer) before study drug administration.
13. Subject has a positive screen for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 and 2 antigens/antibodies.
14. Subject has had a clinically significant acute illness within 4 weeks or other illness within 5 days before the first study drug administration.
15. Subject or a family member of the subject is a member of the professional or ancillary personnel working at the investigative site involved in the study.
16. Not suitable for entry into the study in the opinion of the Investigator.
17. Receipt of blood products within 2 months prior to Check-in.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Part A, B, C, D and E: Incidence and severity of Adverse Events | Up to 28 days after last administration
  A treatment-emergent adverse events (TEAE) will be summarized by treatment and overall, and summarized for each treatment by severity and relationship to study drug. All TEAEs leading to withdrawal, or SAEs, will be summarized.
Part A, B, C, D and E: Number of subjects with clinical laboratory test abnormalities | Up to 28 days after last administration
  The clinical laboratory will include hematology (hematocrit, hemoglobin, mean cell hemoglobin, mean cell hemoglobin concentration, mean cell volume, platelet count, red blood cell count, white blood cell count), clinical chemistry (alanine aminotransferase, albumin, alkaline phosphatase, aspartate aminotransferase, blood urea nitrogen, calcium, chloride, cholesterol, creatinine, creatine phosphokinase, direct bilirubin, estimated glomerular filtration rate, gamma glutamyl transferase, glucose. inorganic phosphate, iron, lactate dehydrogenase, phosphorus, potassium, sodium, total bilirubin, total CO2, total protein, triglyceride, urea, uric acid), and urinalysis (bilirubin, blood, color and appearance, glucose, ketones, leukocyte esterase, nitrite, pH, protein, specific gravity, urobilinogen, microscopic examination, electrolytes). Abnormality will be determined by the investigator.
Part A, B, C, D and E: Number of subjects with vital signs abnormalities | Up to 28 days after last administration
  The vital sign will include blood pressure (mmHg), pulse rate (bpm), respiratory rate (breaths/min), and body temperature (degree Celsius). Abnormality will be determined by the investigator.
Part A, B, C, D and E: Number of subjects with clinically significant change in body weight | Up to 28 days after last administration
  Change in body weight (kg) at baseline and post dose will be measured. Clinical significance will be determined by the investigator.
Part A, B, C, D and E: Number of subjects with abnormal findings in physical examinations | Up to 28 days after last administration
  The physical examination will typically include general appearance, head and neck, eyes, ear, nose and throat, lymph nodes, thyroid, cardiovascular, respiratory, abdomen, nervous, skin, musculoskeletal, peripheral vascular and extremities and be performed at Investigator's discretion based on reported symptoms. Abnormality will be determined by the investigator.

SECONDARY OUTCOMES:
Part A: AUC0-inf of K-755 | Up to 28 days after single administration
  Area under the plasma concentration-time curve (AUC) from time zero extrapolated to infinity
Part A: AUC0-tlast of K-755 | Up to 28 days after single administration
  AUC from time zero to the time of the last measurable concentration
Part A: Cmax of K-755 | Up to 28 days after single administration
  Maximum plasma concentration
Part A: Tmax of K-755 | Up to 28 days after single administration
  Time of the observed maximum plasma concentration
Part A: t1/2 of K-755 | Up to 28 days after single administration
  Terminal plasma elimination half-life
Part B: AUC0-τ of K-755 | Up to 28 days after repeated administration
  AUC over the dosing interval
Part B: Cmax of K-755 | Up to 28 days after repeated administration
  Maximum plasma concentration
Part B: Tmax of K-755 | Up to 28 days after repeated administration
  Time of the observed maximum plasma concentration
Part B: t1/2 of K-755 | Up to 28 days after repeated administration
  Terminal plasma elimination half-life
Part C: AUC0-inf of K-755 | Up to 14 days after single administration
  Area under the plasma concentration-time curve (AUC) from time zero extrapolated to infinity
Part C: AUC0-tlast of K-755 | Up to 14 days after single administration
  AUC from time zero to the time of the last measurable concentration
Part C: Cmax of K-755 | Up to 14 days after single administration
  Maximum plasma concentration
Part C: Tmax of K-755 | Up to 14 days after single administration
  Time of the observed maximum plasma concentration
Part C: t1/2 of K-755 | Up to 14 days after single administration
  Terminal plasma elimination half-life
Part D: AUC0-inf of K-755 | Up to 14 days after single administration
  Area under the plasma concentration-time curve (AUC) from time zero extrapolated to infinity
Part D: AUC0-tlast of K-755 | Up to 14 days after single administration
  AUC from time zero to the time of the last measurable concentration
Part D: Cmax of K-755 | Up to 14 days after single administration
  Maximum plasma concentration
Part D: Tmax of K-755 | Up to 14 days after single administration
  Time of the observed maximum plasma concentration
Part D: t1/2 of K-755 | Up to 14 days after single administration
  Terminal plasma elimination half-life
Part E: AUC0-τ of K-755 | Up to 14 days after single administration
  AUC over the dosing interval
Part E: Cmax of K-755 | Up to 14 days after single administration
  Maximum plasma concentration
Part E: Tmax of K-755 | Up to 14 days after single administration
  Time of the observed maximum plasma concentration
Part E: t1/2 of K-755 | Up to 14 days after single administration
  Terminal plasma elimination half-life

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX, Clinical Research Pty Ltd, Adelaide, South Australia, Australia